CLINICAL TRIAL: NCT03002324
Title: Tailoring of Vaccine-Focused Messages: Moral Foundations and Disease Salience - Part 2
Brief Title: Tailoring of Vaccine-Focused Messages: Disease Salience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Saad B. Omer, MBBS, MPH, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00087211a
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Human Papillomavirus
Keywords: Vaccines; Childhood Vaccination; Decision Making; Health Belief Model
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Current CDC Message Arm (Active Comparator): Participants randomized to this arm will receive a message developed to directly follow the current message on the CDC's website.
  Interventions: Behavioral: Baseline Survey; Behavioral: Current CDC Message; Behavioral: Post-Intervention Survey
- Cervical Cancer Message Arm (Experimental): Participants randomized to this arm will receive a message focused on cervical cancer risks and prevention and framed to highlight perceived susceptibility, perceived benefit, and self-efficacy.
  Interventions: Behavioral: Baseline Survey; Behavioral: Cervical Cancer Message; Behavioral: Post-Intervention Survey
- Control Message (Sham Comparator): Participants randomized to the control arm will be provided with a short message about the costs and benefits of bird feeding.
  Interventions: Behavioral: Baseline Survey; Behavioral: Control Message; Behavioral: Post-Intervention Survey

INTERVENTIONS:
Behavioral: Baseline Survey — The baseline survey is a combination of the Vaccine Confidence Scale, and a short form of the Parents' Attitudes about Childhood Vaccines (PACV) Scale. Participants will be asked an additional 10 questions developed as a part of a behavioral phenotyping questionnaire to assess behavioral biases at baseline within the study population. Demographic information and intent to vaccinate will also be collected.
Behavioral: Current CDC Message — Participants randomized to the current CDC message arm will read a message taken almost directly from the CDC Vaccine Information Sheet (VIS) on HPV. This message was minimally altered for length and clarity.
  Arms: Current CDC Message Arm
Behavioral: Cervical Cancer Message — Participants randomized to the cervical cancer messaging arm will receive a message developed by the study team to appeal tenants of the Health Belief Model (self-efficacy, perceived benefit) and on the purity tenant of the moral foundations theory.
  Arms: Cervical Cancer Message Arm
Behavioral: Control Message — Participants randomized to the non-vaccine related control arm will read a bird-feeding passage.
  Arms: Control Message
Behavioral: Post-Intervention Survey — The immediate post-intervention survey will include questions from the Vaccine Confidence Scale and the PACV short scale. Intent to vaccinate will be assessed.

SUMMARY:
This study is the second phase of a trial examining decision making about vaccines. For this phase of this study, the researchers will conduct a 3-arm randomized trial to compare the current Centers for Disease Control and Prevention (CDC) human papillomavirus (HPV) message, a new cervical cancer focused message developed by the study team, and a non-vaccine related control passage among parents of adolescent females. The goal of the trial will be to determine if the new cervical cancer framed message has an increased impact on intent to have daughters receive the HPV vaccine over the trial period as compared to the current CDC message used in the field. Additionally, the researchers will examine the impact both the CDC message and the new message individually have on intent to vaccinate when compared to the non-vaccine related control message.

The participant's vaccine beliefs and intent to vaccinate will be assessed through an online survey at baseline. Two weeks later, participants will be randomized to view one of the three messages: the current CDC message, the cervical cancer framed message, or a non-vaccine related control message. Immediately afterwards, vaccine beliefs and intent to vaccinate will be assessed to determine the impact of the message.

DETAILED DESCRIPTION:
Genital human papillomavirus (HPV) is the most common sexually transmitted infection in the United States. Most HPV infections are asymptomatic and clear on their own within 2 years but persistent infections can lead to diseases, including several cancers. Cervical cancer is the most common cancer caused by HPV infection, and virtually all cervical cancers can be attributed to HPV infection. There is no cure for HPV, but HPV can be prevented through vaccination. Current recommendations from the Advisory Committee on Immunization Practices (ACIP) state that the HPV vaccine may be given starting at 11-12 years of age for boys and girls, through age 26. Despite the safety and efficacy of this vaccine, the coverage among adolescents aged 11-17 years old remains low. Attaining high vaccination rates among adolescents is essential to decreasing the burden of disease due to cervical cancer, and other cancers caused by HPV.

Parental decision to vaccinate their children, specifically with the HPV vaccine, can be tied to multiple constructs of the Health Belief Model. These include perceived susceptibility of HPV infection (is my child at risk of infection), perceived benefit, and perceived severity (of disease, and of vaccine related adverse events). This would suggest that messaging surrounding the HPV vaccination should be highly salient within these constructs. The current message tied to the HPV vaccine presented by the Centers for Disease Control (CDC) has a focus on HPV as an infection and is clinical in nature. In a randomized trial, parents given information about HPV were no more likely to be accepting of an HPV vaccine and no more likely to get their child vaccinated. Based on this literature, the researchers hypothesize that reframing the message to promote HPV vaccination as a means of protection against cervical cancer will impact intent to vaccinate among parents of adolescent females (aged 11-17 years old).

In the first phase of this study the researchers assessed how appealing to different moral foundations impacted attitudes towards vaccination and intent to vaccinate. For this phase of this study, the researchers will conduct a 3-arm randomized trial to compare the current CDC HPV, a cervical cancer focused message developed by the study team, and a non-vaccine related control passage among parents of adolescent females. The goal of the trial will be to determine if the new cervical cancer framed message has an increased impact on intent to have daughters receive the HPV vaccine over the trial period as compared to the current CDC message. Additionally, the researchers will examine the impact both the CDC message and the new message have on intent to vaccinate when compared to the non-vaccine related control message.

The participant's vaccine beliefs and intent to vaccinate will be assessed through an online survey at baseline. Two weeks later, participants will be randomized to view one of the three messages: the current CDC message, the cervical cancer framed message, or a non-vaccine related control message. Immediately afterwards, vaccine beliefs and intent to vaccinate will be assessed to determine the impact of the message.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one daughter between 9 and 17 years of age (inclusive)
* Reside in the United States

Exclusion Criteria:

* Have previously participated in the disease salience phase of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1320 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Overall change in attitude towards the human papilloma virus (HPV) vaccine | Week 2
  Number of caregivers experiencing a change in attitude towards the HPV vaccine
Intent to have their child vaccinated against HPV | Week 2
  Number of caregivers intending to have their daughter(s) receive the HPV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Saad B Omer, BBS, MPH, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter RM, Amin AB, Bednarczyk RA, Omer SB. Cancer-salient messaging for Human Papillomavirus vaccine uptake: A randomized controlled trial. Vaccine. 2018 Apr 25;36(18):2494-2500. doi: 10.1016/j.vaccine.2018.01.040. Epub 2018 Mar 26. PMID 29599089